CLINICAL TRIAL: NCT03925766
Title: Laparoscopy-Assisted Transgastric Endoscopic Retrograde Cholangiopancreatography for Choledocholithiasis After Roux-en-Y Gastric Bypass
Brief Title: Laparoscopy-Assisted Transgastric ERCP
Status: Completed | Type: Observational
Sponsor: Tecnologico de Monterrey (Other)
Responsible Party: Sponsor
Other Study IDs: LAERCP002
Record Dates: First submitted 2019-04-22; First posted 2019-04-24 (Actual); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Biliary Obstruction
Keywords: biliary disease; gallstones; obesity
MeSH Terms: conditions — Gallbladder Diseases; Gallstones; Obesity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
We describe a case of a 57-year-old patient with altered RYGB anatomy, who underwent a laparoscopic cholecystectomy with a intra-operative cholangiogram showing a stone on the common bile duct. A laparoscopic assisted trans-gastric ERCP was successfully performed. The presentation of the case is presented as well a review of the literature.

DETAILED DESCRIPTION:
The exclusion of the stomach after Roux-en-Y-Gastric bypass (RYGB) makes access to the biliary tree very challenging for the surgeon or the endoscopist. There are different techniques described to overcome this downside, being laparoscopic assisted trans-gastric endoscopic retrograde cholangiopancreatography (ERCP) approach an outstanding method to access the remnant stomach for reaching the duodenal papilla, with a high rate of success reported. We describe a case of a 57-year-old patient with altered RYGB anatomy, who underwent a laparoscopic cholecystectomy with a intra-operative cholangiogram showing a stone on the common bile duct. A laparoscopic assisted trans-gastric ERCP was successfully performed, introducing the duodenoscope through a gastrostomy without the need of an intra-gastric trocar. The patient evolved favorably and was discharged on his second postoperative day without complications.

ELIGIBILITY:
Inclusion Criteria:

* Patient with altered Roux en Y Gastric Bypass anatomy

Exclusion Criteria:

* Patients without Roux en Y Gastric Bypass anatomy

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with altered Roux en Y Gastric Bypass anatomy
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-20 (Actual)

PRIMARY OUTCOMES:
Proof the efficacy of laparoscopic assisted transgastric endoscopic retrograde cholangiopancreatography | April 2019
  This technique is a feasible and achievable procedure with low rate of complications for treating patients with altered RYGB anatomy that present biliary tract disorders, allowing an endoscopic treatment and cholecystectomy to be performed in a single setting.

CONTACTS AND LOCATIONS:
Locations (1):
- Escuela Nacional de Medicina, Tecnologico de Monterrey, Monterrey, Nuevo León, Mexico